CLINICAL TRIAL: NCT03206957
Title: Interventional Controlled Cross-sectional Study Assessing the Correlation Between Optic Nerve Vessels Anomalies, Serum Angiogenic Factors and Renal Anomalies in Children With Down Syndrome.
Brief Title: Correlation Between Optic Nerve Vessel Anomalies, Serum Angiogenic Factors and Renal Anomalies in Down Syndrome Children
Acronym: DOPANUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P2017/Ophtalmo/DOPANUR
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Urinalysis

STUDY DESIGN:
Intervention Model Description: Interventional controlled cross-sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study group (Other): Down Syndrome children
  Interventions: Diagnostic Test: Funduscopic examination and retinal photography; Diagnostic Test: Serum levels of endostatin and angiogenesis factors; Diagnostic Test: Renal and low urinary tract Doppler ultrasound; Diagnostic Test: Urinalysis; Diagnostic Test: Anthropometric measures and vitals signs
- Control group n°1 (Other): Down Syndrome children's mothers
  Interventions: Diagnostic Test: Funduscopic examination and retinal photography; Diagnostic Test: Serum levels of endostatin and angiogenesis factors
- Control group n°2 (Other): Age and sex matched healthy children
  Interventions: Diagnostic Test: Funduscopic examination and retinal photography; Diagnostic Test: Renal and low urinary tract Doppler ultrasound; Diagnostic Test: Urinalysis; Diagnostic Test: Anthropometric measures and vitals signs
- Control group n°3 (Other): Down syndrome children's healthy siblings
  Interventions: Diagnostic Test: Funduscopic examination and retinal photography; Diagnostic Test: Serum levels of endostatin and angiogenesis factors

INTERVENTIONS:
Diagnostic Test: Funduscopic examination and retinal photography — A standardized funduscopic examination and retinal photography will be performed by an ophthalmologist focusing on optic nerve.
Diagnostic Test: Serum levels of endostatin and angiogenesis factors — Serum levels of endostatin, angiopoietin and vaso endothelial growth factor will be analyzed
  Arms: Control group n°1; Control group n°3; Study group
Diagnostic Test: Renal and low urinary tract Doppler ultrasound — Measurements of each kidney will include maximum renal bipolar length in a sagittal plane, renal width and thickness in an axial plane perpendicular to each other at the level of renal hilum and cortical thickness. Intensity of corticomedullary differentiation will estimated.
  Doppler ultrasound examination will assess renal arterial resistivity indexes
  Arms: Control group n°2; Study group
Diagnostic Test: Urinalysis — Urinalysis assessments will include assessments of microalbuminuria and microalbuminuria to creatinuria ratio. A spot urine sample will be collected from first morning void.
  Arms: Control group n°2; Study group
Diagnostic Test: Anthropometric measures and vitals signs — weight, height and blood pressure will be assessed
  Arms: Control group n°2; Study group

SUMMARY:
In approximately half of individuals with Down syndrome, an higher than normal number of vessels cross the optic disc margin. Investigator hypothesize that early retinal vessel branching occurs due to inhibition of angiogenesis by triplet overexpression of endostatin, an angiogenesis inhibitor encoded on chromosome 21. Since angiogenesis is critical in the development of eyes and other organs angiogenesis depended (specially kidney, brain, and recently described lungs and heart), early branching of retinal vessels at the level of the optic disc would also likely result in abnormal renal and other organs development in these individuals. Investigator wish to determine whether observation of optic disc vessels may serve as an indicator of elevated endostatin levels and other angiogenesis-dependent organs anomalies.

DETAILED DESCRIPTION:
Investigator will measure the serum levels of endostatin as well as others angiogenetic factors in Down syndrome children versus control group 1 constituted by the patient mothers.

Investigator will also perform renal and low urinary tract Doppler ultrasound with measurement of renal dimension in order to determine if the kidneys of patients with high level of serum of endostatin are smaller than those of patients with normal level of endostatin. Data observed in Down syndrome children will be compared to control group 2age constituted by sex and age matched healthy children Urine microalbuminuria and urine microalbuminuria/creatinuria from the first urine in the morning will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Provision of personally signed and dated informed consent document by adult subject or parents
* When capable of providing assent, provision of personally signed and dated informed assent document by children
* Subjects and/or their caregivers/parents are willing and able to comply with scheduled laboratory tests, and other required study procedures.

Exclusion Criteria:

• Inability to cooperate with study related examination

For "Study Group" subjects

* Known chronic diseases unrelated to their triallelic condition For "Control Group n°1" & "Control Group n°3"
* General disease in which the level of endostatin may be modified such as leukemia, cancers, inflammatory diseases (e.g.: rheumatoid arthritis, Crohn's disease, psoriasis)
* Any condition that may cause a hypoxia
* Pregnancy

For "Control Group n°2":

* Healthy children except benign ophthalmological refraction anomalies
* Any known renal or low urinary tract diseases.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between the number of retinal vessels crossing the optic disc and serum level of endostatin | 18 months
  correlation coefficent

SECONDARY OUTCOMES:
Correlation between the number of retinal vessels crossing the optic disc and serum level of other angiogenic factors | 18 months
  correlation coefficent
Correlation between serum level of endostatin and serum level of other angiogenic factors | 18 months
  correlation coefficient
Description of renal anomalies in Down syndrome. | 18 months
  absolute number and type of renal anomalies
Comparison of prevalence of renal anomalies between Down syndrome and healthy subjects | 18 months
  Proportion and type of disease
Correlation between the number of optic nerve vessels and the presence of organs pathologies | 18 months
  correlation coefficient
Correlation between serum level of angiogenesis factors and the presence of organs pathologies | 18 months
  correlation coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Lavina Postolache, MD, Principal Investigator — Queen Fabiola Children's University Hospital
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No